CLINICAL TRIAL: NCT00689286
Title: BION Implantable Microstimulator System
Brief Title: BION Treatment of Knee Osteoarthritis
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Gerald E. Loeb, M.D., Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BT5
Record Dates: First submitted 2008-05-29; First posted 2008-06-03 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-06

CONDITIONS: Osteoarthritis, Knee
Keywords: Knee Osteoarthritis; Neuromuscular stimulator
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- BION "twitch" stimulation (Experimental): The first group will have a stimulation paradigm like that used in a previous feasibility study that preceded the proposed trial, using low-frequency (1-5 PPS) "twitch" stimulation.
  Interventions: Device: BION
- BION tetanic-frequency stimulation (Experimental): The second group will have a stimulation paradigm in which tetanic-frequency stimulation (25-50 PPS) is used to produce fused muscle contractions.
  Interventions: Device: BION
- Standardized program (No Intervention): A third group of experimental subjects will have a standardized program of voluntary exercise.

INTERVENTIONS:
Device: BION — They will be divided into three groups. Two groups of experimental subjects will receive stimulation using BIONs. The first group will have a stimulation paradigm like that used in a previous feasibility study that preceded the proposed trial, using low-frequency (1-5 PPS) "twitch" stimulation. The second group will have a stimulation paradigm in which tetanic-frequency stimulation (25-50 PPS) is used to produce fused muscle contractions. A third group of experimental subjects will have a standardized program of voluntary exercise.
  In Groups 1 and 2, the femoral nerve will be stimulated electrically according to the assigned protocol during the 12 week experimental period after implantation of the devices. Individuals assigned to Group 3, receiving conventional exercise therapy for 12 weeks, will be allowed to receive BIONs at the end of the trial, providing they request BION therapy and they have been at least minimally compliant with the exercises.
  Arms: BION "twitch" stimulation; BION tetanic-frequency stimulation

SUMMARY:
Osteoarthritic changes in the knee are a common cause of pain that restricts the subject's ability to move and may lead to surgical intervention with total knee replacement. Quadriceps muscle strengthening has been shown to improve the dynamic stability of the knee, decreasing pain during locomotion and increasing knee function. However, the gains associated with improved quadriceps strength have been difficult to achieve on a routine clinical basis because the currently available ways to increase muscle strength- through voluntary exercise or surface electrical stimulation- have significant practical problems that limit their use. The aim of this prospective study is to evaluate the safety and effectiveness of neuromuscular stimulation using implantable microstimulators called BIONs to improve the strength, range of motion, and health of the knee in patients with knee osteoarthritis. This investigation is expected to last 12 weeks for each study participant; the trial will be completed over a 3-year period. Patients recruited into the study will have advanced knee osteoarthritis for which total knee replacement surgery is being considered. The proposed study extends a feasibility study carried out in Milan, Italy on five patients with knee osteoarthritis, who were implanted with BIONs.

DETAILED DESCRIPTION:
Knee Osteoarthritis is a common problem with people over the age of 50 and is often debilitating because of the challenges it poses to normal walking function. Research has shown that exercise can lessen the effect of the osteoarthritis in the knee if done diligently. BION®s implanted in the thigh can produce contractions of the quadriceps muscles without much movement of the knee joint, an advantage if moving the knee is painful. In this study, teh subjects will be divided into three groups. Two groups of experimental subjects will receive stimulation using BIONs. The first group will have a stimulation paradigm like that used in a previous feasibility study that preceded the proposed trial, using low-frequency (1-5 PPS) "twitch" stimulation. The second group will have a stimulation paradigm in which tetanic-frequency stimulation (25-50 PPS) is used to produce fused muscle contractions. A third group of experimental subjects will have a standardized program of voluntary exercise.. In Groups 1 and 2, the femoral nerve will be stimulated electrically according to the assigned protocol during the 12 week experimental period after implantation of the devices. Individuals assigned to Group 3, receiving conventional exercise therapy for 12 weeks, will be allowed to receive BIONs at the end of the trial, providing they request BION therapy and they have been at least minimally compliant with the exercises. All participants will be eligible to continue treatment following the initial 12 weeks if medically appropriate and resources permit.

ELIGIBILITY:
Inclusion Criteria:

1. Subject presents with osteoarthritis of the knee with severity defined as Kellgren-Lawrence grade 3-4.
2. Subject is between 18 and 75 years old.
3. Attending physician considers the subject in general good health (other than knee joint osteoarthritis).
4. Subject is mentally capable of understanding the goals and the application of therapy.
5. Subject is able to apply the therapy (with or without help) in the home setting.
6. Subject is willing and capable of giving informed consent.
7. Subject is willing and capable of traveling to testing center at the schedule described above and detailed in Table 2.

Exclusion Criteria:

1. Subject is pregnant, nursing, or planning to become pregnant in the next 12 months.
2. Subject has an electronic implant (e.g. cardiac pacemaker, etc.).
3. Subject has metallic implant (e.g. plates, hip joints) in the buttock or upper leg.
4. Subject has a history of falling.
5. Subject has medical conditions other than OA affecting the legs that could affect treatment or mobility.
6. Subject is 40% or more above the ideal weight recommended by Metropolitan Life.
7. Subject has cancer.
8. Subject is currently enrolled in another clinical trial or research study that involves therapy or intervention which would affect lower extremity mobility.
9. Subject has bilateral knee osteoarthritis.
10. Subject is taking pain medications with dosage not stable for one month.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-04; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
quadriceps isometric strength | pre-exercise, 4w, 8w, 12w

SECONDARY OUTCOMES:
Gait velocity Gait endurance Pain WOMAC | pre-exercise, 8w, 12w

CONTACTS AND LOCATIONS:
Overall Officials: Lucinda Baker, Ph.D, Principal Investigator — University of Southern California
Locations (1):
- USC University Hospital, Los Angeles, California, United States

REFERENCES:
- [Background] Loeb GE, Richmond FJ, Baker LL. The BION devices: injectable interfaces with peripheral nerves and muscles. Neurosurg Focus. 2006 May 15;20(5):E2. doi: 10.3171/foc.2006.20.5.3. PMID 16711659